CLINICAL TRIAL: NCT01382329
Title: A Blinded, Randomized Phase 2/3 Study to Assess Immunogenicity and Safety of Two Different Dose Levels of a Vero Cell-Derived Whole Virus H5N1 Influenza Vaccine in a Healthy Japanese Adult Population Aged 18 to 59 Years
Brief Title: H5N1 Vaccine Study in Japanese Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: Baxter Innovations GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 811001
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2012-09

CONDITIONS: H5N1 Influenza
Keywords: Prophylaxis of influenza infection caused by a pandemic influenza virus (H5N1)
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment group I / Intramuscular (Experimental): 85 subjects to receive 2 intramuscular vaccinations at Dose A on Days 1 and 22
  Interventions: Biological: H5N1 (pre-)pandemic influenza vaccine (whole virion, Vero Cell derived, inactivated)
- Treatment group II / Intramuscular (Experimental): 85 subjects to receive 2 intramuscular vaccinations at Dose B on Days 1 and 22
  Interventions: Biological: H5N1 (pre-)pandemic influenza vaccine (whole virion, Vero Cell derived, inactivated)
- Treatment group III / Subcutaneous (Experimental): 85 subjects to receive 2 subcutaneous vaccinations at Dose A on Days 1 and 22
  Interventions: Biological: H5N1 (pre-)pandemic influenza vaccine (whole virion, Vero Cell derived, inactivated)
- Treatment group IV / Subcutaneous (Experimental): 85 subjects to receive 2 subcutaneous vaccinations at Dose B on Days 1 and 22
  Interventions: Biological: H5N1 (pre-)pandemic influenza vaccine (whole virion, Vero Cell derived, inactivated)

INTERVENTIONS:
Biological: H5N1 (pre-)pandemic influenza vaccine (whole virion, Vero Cell derived, inactivated) — Intramuscular injection into the musculus deltoideus or subcutaneous injection in the upper arm

SUMMARY:
The purpose of this study is to obtain immunogenicity and safety data of two different dose levels of an H5N1 pandemic influenza vaccine in a healthy Japanese adult population aged 18 to 59 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 59 years old at the time of screening
* Subject is generally healthy, as determined by the investigator´s clinical judgement through collection of medical history and performance of a physical examination
* Subject is physically and mentally capable of participating in the study and willing to adhere to study procedures to include completion of all elements of the study diary
* If female of childbearing potential, subject presents with a negative urine pregnancy test result within 24 hours prior ot the scheduled first vaccination and agrees to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Subject has a history of infectin with H5N1 virus or a history of vaccination with an H5N1 influenza vaccine
* Subject is at high risk of contracting H5N1 influenza infection (e.g. poultry workers)
* Subject currently has or has a history of a significant cardiovascular (including hypertension), respiratory (including asthma), metabolic, neurological (including Guillain-Barré Syndrome and acute disseminated encephalomyelitis), hepatic, rheumatic, autoimmune, hematological, gastrointestinal or renal disorder
* Subject has any inherited or acquired immunodeficiency
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to: systemic or inhaled corticosteroids, radiation treatment, or other immunosuppressive or cytotoxic drugs
* Subject has a history of severe allergic reactions or anaphylaxis
* Subject has a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating
* Subject has received a blood transfusion or immunoglobulins within 90 days prior to study entry
* Subject has donated blood or plasma within 30 days prior to study entry
* Subject has received any influenza or any live vaccine within 4 weeks or any other inactivated vaccine within 2 weeks prior to vaccination in this study
* Subject has a functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse
* Subject was administered an investigational drug within 6 weeks prior to study entry or is concurrently participating in a clinical study that includes the administration of an investigational product
* Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator/subinvestigator or site personnel conducting the study
* If female, subject is pregnant or lactating at the time of enrollment
* Subject has any other condition that disqualifies his/her participation in the study in the opinion of the investigator

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with antibody response to the vaccine strain | 21 days after 2nd vaccination
  Measurement by single radial hemolysis (SRH) assay
Number of subjects demonstrating seroconversion | 21 days after 2nd vaccination
  Measurement by SRH assay
Fold increase of antibody response | 21 days after 2nd vaccination
  Measurement by SRH assay

SECONDARY OUTCOMES:
Number of subjects with antibody response to the vaccine strain | 21 days after 1st and 21+180 days after 2nd vaccination
  Measurement by SRH (except at 21 days after 2nd vaccination), microneutralization (MN) and hemagglutination inhibition (HI) assay
Number of subjects demonstrating seroconversion | 21 days after 1st and 21+180 days after 2nd vaccination
  Measurement by SRH (except at 21 days after 2nd vaccination), MN and HI assay
Antibody response | 21 days after 1st and 21 + 180 days after 2nd vaccination
  Measurement by SRH, MN and HI assay
Fold increase of antibody response | 21 days after 1st and 21+180 days after 2nd vaccination as compared to baseline
  Measurement by SRH (except at 21 days after 2nd vaccination), MN and HI assay

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Geisberger, MD, Study Director — Baxter Innovations GmbH
Locations (3):
- Japan (3):
  - Medical Co. LTA PS Clinic, Fukuoka, Fukuoka
  - CPC Clinic, Medipolis Medical Research Institute, Kagoshima, Kagoshima-ken
  - Osaka Pharmacology Clinical Research Hospital, Osaka, Osaka